CLINICAL TRIAL: NCT03636048
Title: Comparison of General Anesthesia and Combined Spinal-epidural Anesthesia on Postoperative Outcomes in Patients Undergoing Transabdominal Cervico Isthmic Cerclage (TCIC)
Brief Title: Comparison of Anesthesia Type in Patients Undergoing Transabdominal Cervico Isthmic Cerclage (TCIC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough participants
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-05-013
Record Dates: First submitted 2018-08-01; First posted 2018-08-17 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-01

CONDITIONS: Cervical Incompetence
MeSH Terms: conditions — Uterine Cervical Incompetence | interventions — Bupivacaine; Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal anesthesia group (Experimental): Spinal anesthesia is used for operation with epidural patient-controlled device for pain control. Bupivacaine Hcl 0.5% Inj. 9-10mg is injected into intrathecal space for anesthesia. 0.2% ropivacaine is used for postoperative pain control with continuous infusion into epidural space.
  Interventions: Drug: Bupivacaine Hcl 0.5% Inj
- General anesthesia group (Active Comparator): General anesthesia is used for operation with wound patient-controlled device for pain control. propofol (10milligram/ML) 1.5-2 mg/ml is used as bolus intravascular injection for induction of anesthesia. 0.5% ropivacaine is used for postoperative pain control with continous infusion through wound catheter.
  Interventions: Drug: Propofol 10 milligram/ML

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.5% Inj — The patients undergo surgery under spinal anesthesia and a catheter would be inserted into epidural space during the procedure. 0.5% bupivacaine is injected into intrathecal space for spinal anesthesia. For pain control, 0.2% ropivacaine is continuously infused into epidural space postoperatively.
  Other Names: Spinal anesthesia with epidural patient-controlled analgesia
  Arms: Spinal anesthesia group
Drug: Propofol 10 milligram/ML — The patients undergo surgery under general anesthesia and a catheter would be inserted to abdominal incision site at the end of the operation. Propofol is used for induction of general anesthesia, and sevoflurane is used for maintenance of anesthesia. At the end of the operation, the surgeon inserts wound catheter in the surgical site and connects wound patient-controlled analgesia device filled with 0.5% ropivacaine.
  Other Names: general anesthesia with wound patient-controlled analgesia
  Arms: General anesthesia group

SUMMARY:
The investigator aimed to compare the effect of anesthesia on overall postoperative outcomes including post-operative pain score and the fetal well-being (heart rate) in patients undergoing transabdominal cervico isthmic cerclage(TCIC). The investigator divided the patients into two groups. The first group was the patients who undergo general anesthesia with postoperative wound patient-controlled analgesia device(PCA) and the second group was the patients who undergo combined spinal-epidural anesthesia(CSE) with postoperative epidural catheter PCA device for pain control.

DETAILED DESCRIPTION:
Transabdominal cervico isthmic cerclage(TCIC) is performed for the pregnants with Incompetent Internal Os of the Cervix(IIOC) to maintain pregnancy. It is the operation that incise the lower abdomen and ligate the cervix in pelvic cavity. In our center, the surgery was conventionally performed under general anesthesia. Also, for pain control, operator has been inserting a catheter into the incision site and connected the wound PCA. In this way, there were some limitations that the wound PCA could only control the somatic pain and there were significant rates of post-operative nausea and vomiting as common complication of general anesthesia. Thus, the investigator planned to conduct combined spinal-epidural anesthesia(CSE) with postoperative pain control with epidural catheter and compare overall postoperative outcomes with conventional general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo TCIC for IIOC and agree to participate in this study.

Exclusion Criteria:

* Hepatic failure
* Chronic kidney disease(>stage III)
* Hypersensitivity, allergic response and/or resistance to drugs used in this study(ex. pethidine, ropivacaine)
* Spinal anesthesia is not possible
* Refuse to participate in the study
* Cannot understand the agreement
* Body weight is under 50 kg or over 100 kg

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Pain score at 24hours after the end of the operation | Assessed by directly asking to the patient, from date of randomization up to postoperative day 3.
  Numerical Rating Score(0-10), 0:no pain, 5:moderate pain, 10:worst pain

SECONDARY OUTCOMES:
Fetal viability on postoperative day 5 | Assessed by ultrasonography, upto postoperative day 5.
  An obstetrician evaluates fetal viability(fetal heart rate) using ultrasonograph.

CONTACTS AND LOCATIONS:
Overall Officials: Eunmi Choi, MD.PhD, Study Chair — Kangnam sungshim hospital
Locations (1):
- Kangnam sungshim hospital, Seoul, South Korea